CLINICAL TRIAL: NCT02917473
Title: Written Advice to Improve Compliance With Early Detection of Melanoma in First-degree Relatives: a Multicenter, Cluster-randomized Intervention Trial to Evaluate the Impact of Specific Incentives and Study Psychological Determinants of Early Melanoma Detection Behavior in First-degree Relatives
Brief Title: Comparison of Two Strategies for Counseling Skin Examination and Sun Protection in First-degree Relatives of Patients With Melanoma
Acronym: FADEMELA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: Institut national de la santé et de la recherche médicale, CIC 1415, TOURS (Unknown); Institut national de la santé et de la recherche médicale, U930,TOURS (Unknown); Institut d'Enseignement à Distance,University Paris - 8 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: INCA14/LM-FADEMELA; 2016-A00186-45 (Registry Identifier: RCB)
Record Dates: First submitted 2016-07-28; First posted 2016-09-28 (Estimated); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Melanoma; Screening
Keywords: Medical skin examination; Skin Self Examination; Sun protection
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Education and counseling as commonly delivered to the patients in clinical practice.
  Brief oral counseling to the patient focusing on sun protection, self-skin examination, medical skin examination, increased risk of melanoma for their first-degree relatives, who should be informed orally by the patients to protect themselves from UV radiation, perform self-skin examination and ask their GP or dermatologist to perform annual skin examination
  Interventions: Behavioral: In-person counseling; Behavioral: Medical skin screening
- Intervention group (Experimental): Education and counseling as commonly delivered to the patients in clinical practice and written advice for their first-degree relatives.
  In addition to oral counseling to the patient, written advice will be provided to patients for their relatives focusing on sun protection, self-skin examination, medical skin examination, increased risk of melanoma for first-degree relatives, who should also be informed orally by the patients to protect themselves from UV radiation, perform self-skin examination and ask their GP or dermatologist to perform annual skin examinations.
  Interventions: Behavioral: In-person counseling; Behavioral: Written advice; Behavioral: Medical skin screening

INTERVENTIONS:
Behavioral: In-person counseling — In-person counseling
  Sun protection
Behavioral: Written advice — Written advice
  Arms: Intervention group
Behavioral: Medical skin screening — Medical skin screening

SUMMARY:
First-degree relatives of patients with melanoma have a greater risk of developing melanoma. Patients are advised orally to inform their first-degree relatives that they should protect their skin from UV radiation and ask for a skin examination from a general practitioner or dermatologist. The study will evaluate the effectiveness of a written sheet in addition to the usual oral counselling to increase acceptance of skin examination by the first-degree relatives. If effective, written counselling provided to the patient for relatives should be recommended and generalized.

DETAILED DESCRIPTION:
Melanoma (MM) is a common cancer affecting 11,000 new cases per year in France and the incidence has tripled in 30 years. It now includes young people, and is responsible for 1600 deaths /year in France. Greater tumor thickness and delayed diagnosis are associated with higher mortality. Prevention and early detection on a large scale in the general population are effective but expensive. First-degree relatives have a greater risk of developing MM. A study carried out in the USA found that a biennial consultation is justified and cost-effective in first-degree relatives of MM patients. The best way to deliver the message of sun protection and screening by a dermatologist, and the reality of behavioural changes induced by counseling and the psychological determinants of adherence to medical skin examination are not fully understood.

A pilot study performed in our center suggested the value of a short written advice provided for participants to give to their relatives to promote sun protection and medical skin examination. The participants reported a significant increase in interest in medical skin examination by their relatives (p=0.006), but the investigators do not know whether the relatives really consulted for examination.

The aim of the multicenter cluster-randomized study is to demonstrate that a higher ratio of relatives will in fact consult their GP or dermatologist for skin examination in the centers randomized to the intervention arm, i.e advice leaflet and usual oral counselling, compared to the centers randomized in the control arm, i.e. usual oral counselling. Participants and their relatives in the intervention group will be asked to undergo psychological tests to identify potential barriers to skin examination and sun protection.

If effective, the investigators expect to improve the written information and to generalize its distribution at national level.

ELIGIBILITY:
Inclusion Criteria:

For Patients:

* Personal history of Stage 0 through IIB melanoma
* At maximum of 12 weeks after surgical treatment of Stage 0 through IIA melanoma
* Have at least one first-degree relative
* Speaking and reading French
* Affiliated to the French Health Insurance system
* Signed non-opposition form at the 1 year consultation

For 1st degree relatives:

* To be 1st degree related to a patient with melanoma
* Speaking and reading French
* 1st degree relatives informed by patients and agreeing to fill out the psychological questionnaires and to the use of their personal data by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Consulting general practitioner or dermatologist | 1 year
  The number of relatives who will have consulted a dermatologist or a general practitioner to perform whole body skin examination

SECONDARY OUTCOMES:
Self-skin examination reported by the relatives | 1 year
  The number of relatives who declare to have performed Self-skin examination.
Sun protection behaviors reported by the relatives | 1 year
  Sun protection behaviours reported by the relatives and assessed by a questionnaire
Barriers to skin examination identified from psychological questionnaires in patients and their relatives | 1 year
  Psychological barriers of patients and their relatives to skin examination evaluated with several questionnaires and scales.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent MACHET, MD-PHD, Study Director — University Hospital, Tours
Locations (9):
- France (9):
  - CHU - ANGERS , Service de Dermatologie, Angers
  - CHRU BREST Hôpital du Morvan, Institut de Cancérologie et d'Hématologie, Brest
  - GH La Rochelle Ré Aunis-Service de Dermatologie, La Rochelle
  - Ch Le Mans, Le Mans
  - CHU NANTES, Service de Dermatologie, Nantes
  - CHU-Poitiers _LA MILETRIE POLE MEDIPOOL-DERMATO-ALLERGOLOGIE, Poitiers
  - CHU -RENNES -Service de Dermatologie-CHU Pontchaillou, Rennes
  - Centre Eugène Marquis -Service d'Oncologie médicale, Rennes
  - University Hospital of Tours, Service de Dermatologie, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Marce D, Le Vilain-Abraham F, Bridou M, Quereux G, Dupuy A, Lesimple T, Le Corre Y, Wierzbicka-Hainaut E, Legoupil D, Celerier P, Maillard H, Machet L, Caille A. Impact of Distribution of a Tip Sheet to Increase Early Detection and Prevention Behavior among First-Degree Relatives of Melanoma Patients: A Randomized Cluster Trial. Cancers (Basel). 2022 Aug 10;14(16):3864. doi: 10.3390/cancers14163864. PMID 36010858